CLINICAL TRIAL: NCT03051399
Title: Clinical Evaluation of the Effects of EpiCor Brand Yeast Fermentate (Made Using Saccharomyces Cerevisiae) on Digestive Comfort, Intestinal Barrier Function and Prebiotic Modulation of the Gut Microbiota.
Brief Title: Clinical Evaluation of the Effects of EpiCor on Digestive Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProDigest (Industry)
Collaborators: University Ghent (Other); Maastricht University (Other); Embria Health Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-PDEMB1/DRUG15-MB1
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Constipation; Gastrointestinal Discomfort
Keywords: Constipation; Gastrointestinal symptoms of discomfort; Quality of life; Saccharomyces cerevisiae; Gut microbiome
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Pilot study performed according to a randomized, double-blind, placebo-controlled parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding was ensured by the fact that both capsules (placebo and EpiCor) were opaque and had an identical appearance and were packed in identical bottles by Embria Health Sciences and were labeled as A or B. A ProDigest staff member not participating in the study labelled all bottles and assigned them to each subject in accordance with the randomization list. All study participants, all members of ProDigest staff involved in the study and the Drug Research Unit Ghent (University Hospital Ghent) that actually performed the study, were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin, 500 mg/day, single serving
  Interventions: Dietary Supplement: Placebo
- EpiCor (Active Comparator): EpiCor, 500 mg/day, single serving
  Interventions: Dietary Supplement: EpiCor

INTERVENTIONS:
Dietary Supplement: Placebo — The participants will be asked to orally ingest one capsule per day (500 mg maltodextrin, single serving), in combination with 200mL water.
  Arms: Placebo
Dietary Supplement: EpiCor — The participants will be asked to orally ingest one capsule per day (500 mg EpiCor, single serving), in combination with 200mL water.
  Arms: EpiCor

SUMMARY:
Previous in vitro studies suggest that EpiCor is well fermented in the colon and has prebiotic potential. The repeated long-term administration of low doses of EpiCor in the Simulator of the Human Intestinal Microbial Ecosystem (SHIME) has shown that this product is able to induce gradual changes in the colonic environment by: i) being selectively fermented, leading to butyrate increase in the colon; ii) stimulating Lactobacilli growth in the lumen and adherence to the mucosal surface, and iii) decreasing potential pathogens. In addition, the fermentation-derived metabolites produced in the colon were shown to potentially benefit the host by decreasing cytokine levels in vitro. As a result, the investigators hypothesize that EpiCor may help to improve bowel function and generally contribute to enhanced gut health. Therefore, this pilot study is intended to assess the effects of long-term administration of EpiCor on a population with mild symptoms of intestinal dysfunction.

The primary objective of this exploratory pilot study is to assess the effect of long term administration of EpiCor on bowel function and gastrointestinal well-being, by means of validated questionnaires.

This study has 4 secondary objectives: 1) The first secondary objective of this study is to assess the protective effects of EpiCor on intestinal barrier function, by performing a gut sugar permeability test in combination with indomethacin challenge; 2) The second secondary objective is to assess the effects of EpiCor on intestinal barrier function, by measuring blood Zonulin and endotoxin levels in combination with indomethacin challenge; 3) The third secondary objective of this study is to assess the prebiotic properties of EpiCor by collecting fecal samples. The microbial community composition, lactate and SCFA profiles and proteolytic activity markers in feces will be determined. Proteolytic activity markers will also be measured in urine samples; 4) The fourth secondary objective of this study is to assess the effects of EpiCor on local and systemic immune system performance by measuring secretory IgA levels in feces and cytokines in blood.

DETAILED DESCRIPTION:
Study design:

In this project the effects of repeated daily intake of EpiCor will be investigated. The design conforms to a randomized, double-blind, placebo-controlled parallel design. In total, there will be two study groups: one group receiving placebo treatment (maltodextrin 500mg daily dose, single serving) and one group receiving EpiCor (500mg daily dose, single serving). Each eligible individual will participate in one of two experimental arms of the study for minimum 6 weeks. Before randomization, there will be a run-in period of 2 weeks in which the participants are prohibited from consuming products containing pre- or probiotics.

Study population:

Healthy human male/female volunteers with mild symptoms of intestinal dysfunction. Subject recruitment will start after ethics committee approval of the study. After obtaining signed informed consent and confirmation of eligibility, each subject will have 4 test days at the study site. Each subject will participate during approximately 8 to 10 weeks in this study. In total, 80 subjects will complete the study (40 subjects in each trial arm). For any patient withdrawn from the study, an alternative candidate will be selected in order to ultimately meet the required number of subjects. The total study duration will be approximately 20 weeks.

Study endpoints:

The primary endpoint for this study is the effect of long-term administration of EpiCor on digestive comfort. Digestive comfort will be assessed by means of evaluation (questionnaires) of i) Gastrointestinal (GI) symptoms (bloating/distension; passage of gas; GI rumbling; feeling of fullness and abdominal discomfort) and ii) frequency/consistency of stools. General gastrointestinal well-being and improvement of quality of life will also be evaluated by means of questionnaires.

Secondary endpoints are i) the protective effects of EpiCor on gut barrier function after indomethacin challenge (assessed by a sugar test in urine samples), ii) the effects of EpiCor on gut barrier function after indomethacin challenge (assessed by quantification of Zonulin in blood), iii) evaluation of EpiCor's prebiotic properties (assessed by microbiota-related analyses on fecal contents) and iv) the effect of EpiCor on local and systemic immune system performance (assessed by measuring secretory (s)IgA levels in feces and cytokines in blood).

Study product:

EpiCor (Embria Health Sciences) is the brand name for a substance consisting of a dried yeast fermentate made using Saccharomyces cerevisiae fermentation. All published human studies on EpiCor used a daily dosage of 500mg for adults. Moreover, this is the commercially recommended daily dosage, and will also be used in this study. The placebo used in this study is Globe maltodextrin 10 (CPIngredientes, Mexico). This commercially available product is a mixture of dextrose, maltose, oligo and polysaccharides obtained by partial enzymatic hydrolysis of corn starch. Maltodextrin is the most commonly used placebo in dietary studies evaluating gut microbiota and intestinal well-being. It is easily digestible and rapidly absorbed as glucose and has no effect on colonic fermentation.

EpiCor and placebo will be provided in capsules. The capsules used in this study will be the Coni-Snap® capsules, two-piece hard gelatin capsules (Capsugel, Mexico).

Blinding procedures:

Blinding is ensured by the fact that both capsules are opaque and have an identical appearance and are packaged in identical bottles by Embria Health Sciences. A ProDigest staff member not participating in the study will label all bottles and assign them to each subject in accordance to the randomization list. The capsules will be packed in identical bottles. Each bottle will contain a weekly dose (=7 capsules per bottle).

The participants will be asked to orally ingest one capsule per day, in combination with 200mL water. The capsules will consist of 500mg EpiCor® or 500mg maltodextrin. To ensure a standardized intake, participants will be asked to take the capsule every morning before breakfast. No interactions with food are reported, and so participants may proceed with their usual food habits. Participants will be asked to hand in the empty bottles; these will be used to measure compliance.

The products are to be stored at room temperature in dry conditions in the closed bottles (preferably between 15 and 25 °C) for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history, healthy volunteers without clinical diagnosed diseases with relevant effect on gastrointestinal system or on visceral motility.
* At the moment of initial inclusion subjects will be recruited for run-in phase if having reported:

  1. Gastrointestinal (GI) symptoms of at least 5 points for the previous 3 months based on self-assessment, or
  2. Reduced bowel movements defined as an average of >1 and ≤5 stools per week for the previous 3 months based on self assessment.
* For at least 50 subjects, an additional inclusion criterion will have to be met based on the daily recorded GI symptoms: at the end of the run-in phase, a score of > or = 5 for GI symptoms should be obtained based on the average calculated from the daily scores of the 2-week run-in period. For the remaining 30 subjects, no additional inclusion criterion will be required.
* Age > or = 18 and < or = 70 years.
* Male or female.
* No pregnancy in the last 6 months.
* Body mass index (BMI) 18-35 kg/m2 (BMI = weight (kg) divided by length (m) squared).
* Consistently stable body weight (± 5%) for at least 6 months and no weight reduction treatment during the study period.
* Written consent to participate in the study.
* Able and willing to follow the study protocol procedures

Exclusion Criteria:

* History of severe gastrointestinal/hepatic, hematological/immunologic, metabolic/nutritional disorders, endocrine disorders, celiac disease, type I diabetes mellitus, major surgery and/or laboratory assessments which might limit participation in or completion of study period. Participants having other diseases will be considered or not for randomization after careful evaluation by the principle investigator.
* Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to first dosing. Some medication may be used, if it is considered not to influence gastrointestinal function and motility, upon mutual agreement of the investigator and sponsor.

  a. In particular, the use of any non-steroidal inflammatory drugs (NSAIDs) starting 14 days prior to first dosing is prohibited.
* Systemic antibiotics treatment within 60 days prior to first dosing.
* Intake of laxatives or anti-diarrheic drugs within 14 days prior to first dosing.
* Change of dietary habits within the 4 weeks prior to screening (for instance start of a diet rich in fibers).
* Participants anticipating a change in lifestyle or physical activity levels during the study.
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 60 days prior to first dosing.
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgment of the principle investigator).
* Known pregnancy or lactation (checked by a pregnancy test before start of study).
* Dependence on illegal drugs or alcohol.
* Smoking within the last 3 months.
* Blood donation within 1 month before study period.
* Prohibited use of pro-, pre- or synbiotics from 30 days before first dosing and during the study period. A list with forbidden products will be provided.
* Hepatitis C-, B- or HIV-positive (to be tested before start of study).
* History of any major side effects towards intake of pro- or prebiotic supplements of any kind.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Symptoms of gastrointestinal discomfort | Daily for 8 weeks
  The volunteers will be asked to document daily (during the 2-week run-in phase and 6-week intervention phase) their Gastrointestinal (GI) symptoms. For assessment of GI symptoms, the volunteers will be asked to grade daily in the evening the average severity over the previous 24 hours on a 5-point scale from 0 (not at all) to 4 (extremely) for the following GI characteristics: bloating/distension, passage of gas, GI rumbling, feeling of fullness and abdominal discomfort. The run-in diary will also be used as an instrument to include/exclude volunteers from the study after proper assessment during the 2 week run-in phase (see additional inclusion criteria).
Stool frequency and consistency | Daily for 8 weeks
  The volunteers will be asked to document daily (during the 2-week run-in phase and 6-week intervention phase) their stool frequency and consistency. Stool consistency will be recorded by using the Bristol Stool Form Scale (watery or mushy, soft blobs, normal sausage, hard shaped sausage, hard lumps).
General gastrointestinal well-being | 3 visits (V1=baseline, V2=3-weeks intervention, V3=6-weeks intervention)
  General gastrointestinal well-being will also be evaluated by means of one additional questionnaire: the Patient Assessment of Constipation Symptoms (PAC-SYM) (Janssen Global Services, LLC, USA). This questionnaire was developed and validated in a patient population with history of chronic constipation. The PAC-SYM questionnaire is a 12-item self-reporting instrument divided into abdominal, rectal, and stool domains, which will be used to assess the constipation symptoms at the beginning (after 2-week run-in phase; visit 1), middle (after 3-weeks intervention; visit 2) and end of intervention (after 6-weeks intervention; visit 3) retrospectively. A 5-point scale from 0 (absent) to 4 (very severe) is used to assess the different symptoms.
Constipation-associated quality of life | 3 visits (V1=baseline, V2=3-weeks intervention, V3=6-weeks intervention)
  Constipation-associated quality of life will also be evaluated by means of one questionnaire: the Patient Assessment of Constipation Quality of Life (PAC-QOL) (Janssen Global Services, LLC, USA). This questionnaire was developed and validated in a patient population with history of chronic constipation. The PAC-QOL provides information about the special distraction of daily life and general well-being of volunteers because of constipation. The PAC-QOL questionnaire is a 28-item self-reporting instrument divided into four domains: physical discomfort, psychosocial discomfort, worries and concerns and satisfaction. This will be filled in by the participants at the same time as PAC-SYM: at the beginning (after 2-week run-in phase; visit 1), middle (after 3-weeks intervention; visit 2) and end of intervention (after 6-weeks intervention; visit 3) retrospectively. A 5-point scale from 0 (none of the time) to 4 (all of the time) is used to assess the different symptoms.
Perceived stress | 3 visits (V1=baseline, V2=3-weeks intervention, V3=6-weeks intervention)
  It is known that psychosocial factors, such as daily stress may alter gut physiology leading to ileum contractions and consequently to GI discomfort. Therefore, subjects will be asked to scale their stress levels in the Perceived Stress Scale (PSS) questionnaire. This is the most widely used psychological (and generic) instrument for measuring the perception of stress. This is a 10-item self-reporting. This will be filled in by the participants at the same time as PAC-SYM and PAC-QOL: at the beginning (after 2-week run-in phase; visit 1), middle (after 3-weeks intervention; visit 2) and end of intervention (after 6-weeks intervention; visit 3) retrospectively. A 5-point scale from 0 (never) to 4 (very often) is used to assess the different symptoms.

SECONDARY OUTCOMES:
Intestinal barrier function: the Multi-Sugar Permeability Test | 2 visits (V1=baseline, V3=6-weeks intervention)
  The first secondary endpoint is to assess the protective effects of EpiCor on intestinal barrier function after indomethacin challenge, by performing a gut sugar permeability test. Indomethacin is able, even after only two doses, to reversibly increase intestinal permeability. Therefore, this test will be performed after the intake of 75 and 50mg of indomethacin on the evening prior to and on the morning before the test, respectively. This test, known as the multi-sugar (MS) test, is performed in urine samples collected for 24 hours after the intake of 5 orally administered sugar probes (sucrose, lactulose, rhamnose, sucralose and erythritol).
Intestinal barrier function: Zonulin and Endotoxin levels | 2 visits (V1=baseline, V3=6-weeks intervention)
  The second secondary objective is to assess the effects of EpiCor on intestinal barrier function, by measuring blood Zonulin and endotoxin levels. Alterations in the integrity of the mucosal barrier are known to be involved in gut inflammatory diseases, obesity and metabolic syndrome. Gut barrier is sustained by tight junction proteins that keep adjacent epithelial cells together, thereby forming a virtually impermeable barrier to fluids. Zonulin is a protein able to modulate the intestinal barrier by disassembling the tight intercellular junctions that characterize the early phase of inflammatory states. Therefore, Zonulin up-regulation is associated with increased permeability. Circulating LPS may be determined in plasma samples in order to assess the effect of the intervention in low-grade endotoxemia.
Prebiotic properties: Gut microbiota analysis | 3 visits (V1=baseline, V2=3-weeks intervention, V3=6-weeks intervention)
  Metabolites' analysis - Lactate, SCFA, BCFA, Ammonia and Enzymatic activity:
  The third secondary objective is to assess the prebiotic properties of EpiCor by collecting fecal samples. The microbial community composition, lactate and short-chain fatty acid (SCFA) profiles in faeces will be determined. Proteolytic activity markers (Branched chain fatty acids - BCFA) in faeces will also be measured
  Microbiota composition and structure:
  Changes in the general composition and structure of the gut microbiome will be studied by sequencing the 16S rRNA region which is common to most prokaryotes. Among the bacteria with known benefits to the host, are the genera Bifidobacterium and Lactobacillus, possibly the two most studied and recognized genera as containing probiotic species. Thus, in addition, quantitative (q)PCR will be done specifically to quantify the relative increase or decrease of these two genera in fecal samples collected after intervention and compare it to baseline.
Immune function | 3 visits (V1=baseline, V2=3-weeks intervention, V3=6-weeks intervention)
  The state of low-grade inflammation elicited by circulating LPS may trigger the expression of inflammatory cytokines. Therefore, the expression of cytokines in blood serum samples will be determined. Secretory IgA (SIgA) is the most abundant class of antibodies found in the intestinal lumen of humans, and is recognized as a first line of defense in protecting the intestinal epithelium from enteric pathogens and toxins. Besides its role in active immune defense, it is also involved in immune tolerance and in maintenance of intestinal homeostasis, by being induced by tolerogenic cytokines such as transforming growth factor beta (TGF-b) and interleukin (IL)-10. Therefore, this is a recognized marker for gut immune regulation, which can be modulated by dietary supplements. Blood serum samples will be used to measure cytokine levels. Fecal samples collected before, during and after intervention will be used to assess the levels of SIgA.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Pinheiro, PhD, Principal Investigator — ProDigest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinheiro I, Robinson L, Verhelst A, Marzorati M, Winkens B, den Abbeele PV, Possemiers S. A yeast fermentate improves gastrointestinal discomfort and constipation by modulation of the gut microbiome: results from a randomized double-blind placebo-controlled pilot trial. BMC Complement Altern Med. 2017 Sep 4;17(1):441. doi: 10.1186/s12906-017-1948-0. PMID 28870194